CLINICAL TRIAL: NCT06765265
Title: Impact of Atorvastatin Versus Rosuvastatin on 25 Hydroxy Vitamin D Levels in Patients With Acute Coronary Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Sidrah Lodhi, Assistant Professor of Endocrinology, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 508/RC/KEMU/13-11-2023
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Coronary Syndromes
Keywords: atorvastatin; rosuvastatin; Vitamin D; Triglyceride; Lipid Profile
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Active Comparator): Atorvatstain 40mg OD
  Interventions: Drug: Atorvastatin 40 mg
- Rosuvastatin (Experimental): Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin 20 mg/day

INTERVENTIONS:
Drug: Rosuvastatin 20 mg/day — Rosuvastatin 20 mg / Day for 24 weeks
  Arms: Rosuvastatin
Drug: Atorvastatin 40 mg — Atorvastatin 40mg / Day for 24 weeks
  Arms: Atorvastatin

SUMMARY:
there will be 2 groups of patients with acute coronary syndrome. The patients will receive one of the 2 study drugs and impact on raising Vitamin D level will be seen after 6 months

DETAILED DESCRIPTION:
this randomized clinical trial will include 152 patients of acute coronary syndrome with normal Vitamin D levels. they will be randomized to receive either Atorvastatin or Rosuvastatin. After 6 months of therapy, the impact on Vitamin D levels will be checked

ELIGIBILITY:
Inclusion Criteria:

Acute Coronary Syndrome

25 OH-Vitamin D levels between 30-70ng/ml

Exclusion Criteria:

Hypercalcemia

hypocalcemia

pregnancy

lactation

hypersensitivity to statins

hypothyroidism

Deranged LFTs & RFTs

Use of following within last 3 months (Vitamin D Supplements, lipid lowering drugs, anti-obesity drugs, corticosteroids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum Vitamin D | 24 weeks

SECONDARY OUTCOMES:
Lipid Profile | 4 weeks & 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Malik, Study Chair — King Edward Medical University; Ali Hussnain, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: January 2025-January 2026

REFERENCES:
- [Result] Althanoon Z, Faisal IM, Ahmad AA, Merkhan MM, Merkhan MM. Pharmacological aspects of statins are relevant to their structural and physicochemical properties. Systematic Reviews in Pharmacy. 2020 Jul 1;11(7):167-71
- [Result] Levinson SS. Non-High-Density Lipoprotein Cholesterol and Guidelines for Cholesterol Lowering in Recent History. Lab Med. 2020 Jan 2;51(1):14-23. doi: 10.1093/labmed/lmz032. PMID 31147695
- [Result] Sathyapalan T, Shepherd J, Arnett C, Coady AM, Kilpatrick ES, Atkin SL. Atorvastatin increases 25-hydroxy vitamin D concentrations in patients with polycystic ovary syndrome. Clin Chem. 2010 Nov;56(11):1696-700. doi: 10.1373/clinchem.2010.144014. Epub 2010 Sep 3. PMID 20817794
- [Result] Thabit A, Alhifany A, Alsheikh R, Namnqani S, Al-Mohammadi A, Elmorsy S, Qari M, Ardawi M. Effect of simvastatin and atorvastatin on serum vitamin d and bone mineral density in hypercholesterolemic patients: a cross-sectional study. J Osteoporos. 2014;2014:468397. doi: 10.1155/2014/468397. Epub 2014 Aug 13. PMID 25197610
- [Result] Anagnostis P, Adamidou F, Slavakis A, Polyzos SA, Selalmatzidou D, Panagiotou A, Athyros VG, Karagiannis A, Kita M. Comparative Effect of Atorvastatin and Rosuvastatin on 25-hydroxy-Vitamin D Levels in Non-diabetic Patients with Dyslipidaemia: A Prospective Randomized Open-label Pilot Study. Open Cardiovasc Med J. 2014 Jul 11;8:55-60. doi: 10.2174/1874192401408010055. eCollection 2014. PMID 25110531
- [Result] Demir CC, Mousa U, Anil C. Effects of atorvastatin and rosuvastatin therapy on serum 25-hydroxyvitamin D levels: A comparative study 13th European Congress of Endocrinology. Endocr Abstr. 2011;26(1):548.
- [Result] Bauddh NK, Ranga GS. A study of the effect of rosuvastatin on vitamin D levels in patients with hypertension, diabetes mellitus, and coronary artery disease. Int J Health Sci Res. 2016; 6(7):42-6
- [Result] Patwardhan VG, Mughal ZM, Padidela R, Chiplonkar SA, Khadilkar VV, Khadilkar AV. To study impact of treatment with Rosuvastatin versus Atorvastatin on 25 hydroxy Vitamin D concentrations among adult Indian men- a randomized control trial. Indian J Pharmacol. 2020 Sep-Oct;52(5):365-371. doi: 10.4103/ijp.IJP_93_18. PMID 33283767
- [Result] Jorge AJ, Cordeiro JR, Rosa ML, Bianchi DB. Vitamin D deficiency and cardiovascular diseases. Int J Cardiovas Sci. 2018;31(1):422-32
- [Result] Sahebkar A, Reiner Z, Simental-Mendia LE, Ferretti G, Della Corte C, Nobili V. Impact of Statin Therapy on Plasma Vitamin D Levels: A Systematic Review and Meta-Analysis. Curr Pharm Des. 2017;23(6):861-869. doi: 10.2174/1381612822666161006150542. PMID 27719645
- [Result] Radhakrishnan A, Ruckmani A, Abishek M, Govindaraju S. Statin therapy and Vitamin D. Int J Basic Clin Pharmacol. 2015;4:1113-7.
- [Result] Bhattacharyya S, Bhattacharyya K, Maitra A. Possible mechanisms of interaction between statins and vitamin D. QJM. 2012 May;105(5):487-91. doi: 10.1093/qjmed/hcs001. Epub 2012 Feb 9. No abstract available. PMID 22323613
- [Result] Scragg R. The Vitamin D Assessment (ViDA) study - Design and main findings. J Steroid Biochem Mol Biol. 2020 Apr;198:105562. doi: 10.1016/j.jsbmb.2019.105562. Epub 2019 Dec 3. PMID 31809866
- [Result] Verdoia M, Pergolini P, Rolla R, Nardin M, Schaffer A, Barbieri L, Daffara V, Marino P, Bellomo G, Suryapranata H, De Luca G; Novara Atherosclerosis Study Group (NAS). Impact of high-dose statins on vitamin D levels and platelet function in patients with coronary artery disease. Thromb Res. 2017 Feb;150:90-95. doi: 10.1016/j.thromres.2016.12.019. Epub 2016 Dec 28. PMID 28068529